CLINICAL TRIAL: NCT02703896
Title: "Effect of Orally Administered Two Successive Doses of PPIs and/ or H2RAs Without or With a Prokinetic Drug, on the Intragastric pH and Volume and Bile Refluxate in Adults Patients Undergoing Elective Surgery.
Brief Title: Prophylaxis for Aspiration of Gastric Contents.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, ALTAF HUSSAIN, Assistant professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-546
Record Dates: First submitted 2016-02-28; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Aspiration of Gastric Contents
Keywords: g a, bile reflux. PPIs, H2RAs, prokinetic agents
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents | interventions — Lansoprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group C (placebo) (Placebo Comparator): Drug intervention Two doses of Placebo at 8.00 pm and then at 6.00 am
  1. Group C (placebo)
  2. Group C (placebo)
  3. Group C (placebo)
  4. Group C (placebo)
  5. Group C (placebo)
  6. Group C (placebo)
  7. Group C (placebo)
  8. Group C (placebo)
  9. Group C (placebo)
  10. Group C (placebo)
  Interventions: Drug: Drug either PPIS or H2RA and prokinetics; Procedure: orogastric intubation
- Either PPIs or H2RAs (Active Comparator): Drug Intervention Two doses at 8.00 pm and then at 6.00 am
  1. Group L (lansoprazole 15 mg)
  2. Group E(esomeprazole 20 mg)
  3. Group P (pantoprazole 20 mg)
  4. Group R (rabeprazole 10 mg)
  5. Group O (omeprazole 20 mg)
  6. Group T (cimetidine 200 mg)
  7. Group F (famotidine 20 mg)
  8. Group N (nizatidine 150 mg)
  9. Group Z (ranitidine 150 mg)
  10. Group S (lafutidine 10 mg)
  Interventions: Drug: Drug either PPIS or H2RA and prokinetics; Procedure: orogastric intubation
- Either PPIs or H2RAs+prokinetics (Active Comparator): Drug intervention Two doses at 8.00 pm and then at 6.00 am
  1. Group L D (lansoprazole 15 mg+ domperidone 10 mg)
  2. Group EM (esomeprazole 20 mg+metoclopramide 10 mg)
  3. Group PD (pantoprazole 20 mg+domperidone 10)
  4. Group RM (rabeprazole 10 mg+metoclopramide 10 mg)
  5. Group OD (omeprazole 20 mg+domperidone 10)
  6. Group TD (cimetidine 200 mg+domperidone 10)
  7. Group FM (famotidine 20 mg+metoclopramide 10 mg)
  8. Group NM (nizatidine 150 mg+metoclopramide 10 mg)
  9. Group ZD (ranitidine 150 mg+ domperidone 10 mg)
  10. Group SD (lafutidine 10 mg+domperidone 10 mg)
  Interventions: Drug: Drug either PPIS or H2RA and prokinetics; Procedure: orogastric intubation
- Either PPIs or H2RAs+Prokinetic (Active Comparator): Drug intervention Two doses at 8.00 pm and then at 6.00 am Group OM (omeprazole 20 mg +metoclopramide 10 mg) Group SM (lafutidine 10 mg + metoclopramide 10 mg )
  Interventions: Drug: Drug either PPIS or H2RA and prokinetics; Procedure: orogastric intubation
- Intervention Orogastric intubation (Other): After general anesthesia, an oro-gastric tube was inserted through another endotracheal tube placed in upper esophagus into the stomach for aspiration of gastric contents.
  Interventions: Drug: Drug either PPIS or H2RA and prokinetics; Procedure: orogastric intubation

INTERVENTIONS:
Drug: Drug either PPIS or H2RA and prokinetics — Drug intervention ( dose unit mg) Two oral doses 8:00 p.m. and 6:00 a.m. (n=60) total 10 groups
  1. Group C (placebo),Group L (lansoprazole15 ), Group LD (Lansoprazole 15 +domperidone 10 )
  2. Group C ,R (rabeprazole 10), RM (rabeprazole 10 + metoclopramide 10)
  3. Group C , E (esomeprazole 20 ), and EM (esomeprazole 20 + metoclopramide 10)
  4. Group C, P (pantoprazole 20), and PD (pantoprazole 20 + domperidone 10 mg)
  5. Group C, O (omeprazole 20), OD (omeprazole 20 + domepridone 10), OM (omeprazole 20 + metoclopramide 10)
  6. Group C,T (cimetidine 200), TD (cimetidine 200 + domperidone 10)
  7. Group C , Z (ranitidine 150), ZD (ranitidine 150 + domperidone 10)
  8. Group C , N (nizatidine 150),NM (nizatidine 150 + metoclopramide 10)
  9. Group C, F (famotidine 20 mg), and FM (famotidine 20 mg + metoclopramide 10)
  10. Group C,S (lafutidine 10), SD (lafutidine 10 + domperidone 10), and Group SM (lafutidine 10 + metoclopramide 10)
  Other Names: Drug treatment; lansoprazole, esomeprazole,pantoprazole,rebeprazole, omeprazole,cimetidine,nizatidine,famotidine,ranitidine,lafutidine
Procedure: orogastric intubation — OGT insertion:Insertion of orogastric tube(through an endotracheal tube placed in the upper esophagus) into the stomach after general anaesthesia.
  Other Names: OGT Insertion

SUMMARY:
Effect of orally administered two equal and consecutive doses of proton pump inhibitors, omeprazole, lansoprazole, esomeprazole , rabeprazole and pantoprazole and Histamine 2 receptor antagonists cimetidine, ranitidine,famotidine,nizatidine and lafutidine without and with a prokinetic agents domperidone, metoclopramide and erythromycin on intragastric pH, volume and bile refluxate.

DETAILED DESCRIPTION:
(This description is for one drug and similar for other drugs) We repacked the placebo, lansoprazole 15 mg and lansoprazole 15 mg plus domperidone 10 mg in 180 envelopes (times two) and then two envelope in one envelope each for evening and morning of the same size, shape and color and their name were changed as drug one, drug two and drug three by a person who was not taking part in the study to the patients (single-blind) and investigators (double-blind) blinded of it. The group assign paper was sealed in another envelope that was opened to know which drug corresponds to either drug one or drug two or drug three after the statistical analysis(triple-blind).

On the preoperative anaesthesia visit, a day before surgery, the nature and purpose of the study was explained to each patient. We asked each patient to pick up on one envelop from the envelopes (randomization). Thus the patients were allocated to either Group C (control), Group L lansoprazole 15 mg or Group LD lansoprazole 15 mg with domperidone 10 mg randomly by sealed envelope method. Age, sex, ASA physical status, weight, height, BMI and the study drug given were recorded for each patient. All patients also received tablet diazepam 5 mg with study drugs. These drugs were given orally with 20 ml of drinking water at 8:00 p.m. in the evening day before surgery and 6:00 a.m. morning on the day of surgery. According to the hospital policy, all patients were fasted from 12:00 midnight. Upon arrival in the receiving area of the operating room. All patients were asked if they had been aware of any unusual feeling (side effect) after taking the study drug.

In the operating room, routine monitors were attached to the patients and turned on. After pre-oxygenation with 100% O2 by face mask using eight breaths vital capacity method, anaesthesia was induced with injection fentanyl 1-2 mcg/kg, propofol 2-3 mg/kg and rocuronium 0.6-0.9 mg/kg. Lungs were ventilated taking care not to inflate the stomach. Maintaining cricoid pressure trachea was intubated with cuffed endotracheal tube. Placement and position was confirmed with EtCO2 monitor and then secured properly. After establishing stable anaesthesia, an endotracheal tube sized 8.5 internal diameter was passed via oral route in the esophagus with anterior displacement of larynx. A predetermined length marked with adhesive tape (xiphoid process to ear lobule- fro ear lobule to nasal tip) of stomach tube sized 18 F was passed through the esophageally placed endotracheal tube. Placement of this tube within the stomach was verified with auscultation over the epigastrium during insufflation of 10-15 ml of air. Gastric contents were gently aspirated manually with 60 ml syringe by an investigator who was blind of group assignment. Applying manual pressure over the epigastrium while the patient was in supine and then left and right lateral positions, gastric tube was then manipulated to ensure maximum emptying of gastric contents. The stomach tube was then removed followed by esophageally placed endotracheal tube. Any problem encountered during inserting or removing the oro-esophageally placed endotracheal tube or gastric tube was also recorded. The volume of gastric contents was measured with graduated syringe and pH using pH meter. The pH meter was calibrated using standard buffers at pH values of 4, 7 and 9.20. This pH meter has a precision of 0.01 units over the entire pH range. A minimum of one-millimeter volume of gastric contents was sufficient for pH determination with pH meter. In case of very little amount of gastric contents, we cut the stomach tube and aspirated gastric material with disposable plastic pipette. Samples less than one-millimeter were considered as no gastric contents because a minimum of one- millimeter of gastric contents was sufficient for pH- metry. Using bile salts as marker for bile, we applied qualitative Hay's sulphur test for the presence of bile salts. A minimum volume of one millimeter of gastric contents was adequate to perform Hay's sulphur test. In this test finely powered sulphur is sprinkled on the surface of cool (17 OC or below) liquid. If bile salts are present sulphur sinks down, sooner or later, in accordance with their percentage. If bile salts are present in from 1:5,000 (0.02%or 200 mcg/ml to 1:10,000 (0.01% or 100 mcg/ml) sulphur at once begins to sink and all precipitated in two or three minutes; even in dilution of 1:120,000 (0.0008% or 8.33 mcg/ml precipitation occurs. On the other hand, if sulphur remains floating on the surface, bile salts are absent.

Anaesthesia was maintained with air, O2 and sevoflorane. Patients also received incremental doses of fentanyl and rocuronium as required. At the end of surgery, injection atropine and neostigmine were given to antagonize the residual effect of rocuronium. All patients were extubated in lateral position and then transferred to recovery room.

Time since premedication T1 (time from evening dose till aspiration of gastric contents) and Time since premedicationT2 (time from morning dose till aspiration of gastric contents), pH, volume of gastric contents and results of Hay's sulphur test were also recorded for all patients.

Statistical test were performed using GraphPad Software, Inc., San Diego, United States and results are expressed as absolute values or mean ± standard deviation SD (SEM). Statistical analysis between the groups were carried out using analysis of variance (ANOVA) for age, BMI, time since premedication T1, time since NPO and T2 , pH and volume. Chi square test was applied for sex, ASA physical status, Hay's test and risk of aspiration according to criteria defined (pH ≤ 2.5 and volume ≥ 0.4ml/kg or 25 ml. Post hoc tests with Bonferrni correction applied where p-value significant(p <0,05). A p-value of less than 0.05 was considered statistically significant. Power analysis revealed that the sample size (n= 30) in each group was of the study was sufficient to detect a difference of 0.7 among the groups in gastric pH and volume at a significant level of 0.05 (=α 0 with a power of 0.85.

ELIGIBILITY:
Inclusion Criteria: ASA I and II aged 15-70 years

-

Exclusion Criteria:

Patients with upper gastrointestinal disorders, Body mass index above 35 kg/m2, Receiving medicines known to effect the secretory and or motor functions of stomach, Had undergone surgery on stomach, With difficult intubation Intestinal obstruction, Partuients and Diabetes

.

-

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1920 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
pH of gastric contents | Immediate after induction of general anaesthesia
  pH was measured with pH meter. Unit whole digit with two decimal point for example, 4.24

SECONDARY OUTCOMES:
volume of gastric contents | Immediate after induction of general anesthesia.
  Measured with graduated syringe. Units milliliters (ml)

OTHER OUTCOMES:
bile salts in the gastric contents | immediate after induction of general anesthesia.
  Hay's Sulfur test performed on gastric contents, reported as positive or negative for bile salts

CONTACTS AND LOCATIONS:
Overall Officials: ALTAF HUSSAIN, FCPS,EDAIC, Principal Investigator — Assistant Professor and Consultant Anaesthetist

IPD SHARING:
Plan to Share IPD: Yes